CLINICAL TRIAL: NCT05342558
Title: Efficacy and Safety of Fluticasone Furoate/Vilanterol vs. Umeclidinium/Vilanterol in Patients With COPD-asthma Phenotype vs. Emphysema Phenotype. A Controled Clinical Trial.
Brief Title: Efficacy and Safety of ICS/LABA vs. LAMA/LABA in Patients With Different COPD Phenotypes.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Respiratory Diseases, Mexico (Other Government)
Responsible Party: Principal Investigator, Alejandra Ramirez Venegas, MD, National Institute of Respiratory Diseases, Mexico
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: C49-17
Record Dates: First submitted 2022-04-05; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: COPD
Keywords: Chronic obstructive pulmonary disease; Biomass; Tobacco; COPD treatment; COPD phenotypes
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fluticasone furoate; GSK573719

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biomass Smoke COPD (Active Comparator): Fluticasone Furoate/Vilanterol 100/25 mcgs. Dry powder inhaler with 30 blisters. 1 inhalation a day for 24 weeks.
  Umeclidinium/Vilanterol 62.5/25 mcgs. Dry powder inhaler with 30 blisters. 1 inhalation a day for 24 weeks.
  Interventions: Drug: Fluticasone Furoate/Vilanterol 100/25 mcgs; Drug: Umeclidinium/Vilanterol 62.5/25 mcgs
- Tobacco Smoke COPD (Active Comparator): Fluticasone Furoate/Vilanterol 100/25 mcgs. Dry powder inhaler with 30 blisters. 1 inhalation a day for 24 weeks.
  Umeclidinium/Vilanterol 62.5/25 mcgs. Dry powder inhaler with 30 blisters. 1 inhalation a day for 24 weeks.
  Interventions: Drug: Fluticasone Furoate/Vilanterol 100/25 mcgs; Drug: Umeclidinium/Vilanterol 62.5/25 mcgs

INTERVENTIONS:
Drug: Fluticasone Furoate/Vilanterol 100/25 mcgs — Dry powder inhaler with 30 blisters. 100/25mcgs a day for 24 weeks.
  Other Names: Relvare
Drug: Umeclidinium/Vilanterol 62.5/25 mcgs — Dry powder inhaler with 30 blisters. 62.5/25mcgs a day for 24 weeks
  Other Names: Anoro

SUMMARY:
This is a randomized, blinded, controlled clinical trial for mexican COPD patients.

Biomass smoke associated COPD (BS-COPD) clinical spectrum is different to the one seen in tobacco smoke associated COPD (TS-COPD). BS-COPD patients present COPD-asthma phenotype or asthma-COPD overlap syndrome (ACOS), TS-COPD patients present mostly the emphysema phenotype. BS-COPD patients have a greater risk of exacerbations in comparison to the emphysema phenotype. Therefore, individualizing treatment in both phenotypes may be very useful among the clinical practitioners.

The investigators expect treatment with FF/V to be superior in preventing COPD exacerbations than the U/V combination in patients with COPD-asthma phenotype; andU/V to be superior than FF/V in patients with the emphysema phenotype.

The general objective of the study is to determine the exacerbations outcome in patients with COPD-asthma vs emphysema phenotype patients, treated with both drugs. Secondary objectives include assessment of pulmonary function tests, quality of life, dyspnea and functional capacity change after a 24 weeks treatment.

DETAILED DESCRIPTION:
Type and duration of the investigation: A randomized, blinded, controlled clinical trial; longitudinal, prospective, 3 years (Sep-2017 through Sep-2020).

Background: COPD associated to biomass smoke (BS-COPD) represents the third of all COPD cases in Latin America, and almost the 2% in general population prevalence studies. BS-COPD clinical spectrum is different to the one seen in COPD associated to tobacco smoke (TS-COPD). While BS-COPD patients present COPD-asthma phenotype or asthma-COPD overlap syndrome (ACOS), TS-COPD patients present mostly the emphysema phenotype.

COPD-asthma phenotype in BS-COPD, probably explains that they have a greater risk of exacerbations in comparison to the emphysema phenotype. Therefore, individualizing treatment in both phenotypes may be very useful among the clinical practitioners, because even though those patients are not included in traditional clinical trials, they are part of every day's practice.

In this sense, providing a specific treatment in this group of patients could change the disease progression, improving symptoms, quality of life, reducing costs, side effects and exacerbations. The investigators hypothesize that COPD-asthma phenotype or asthma-COPD overlap syndrome (ACOS), may get a greater benefit by using a combination LABA/ICS (Fluticasone Furoate/Vilanterol - FF/V) therapy, whereas those with the emphysema phenotype with LABA/LAMA (Umeclidinium/Vilanterol U/V) therapy

The upside of these drugs is that both of them have the same easy-to-use device, and it is inhaled once a day only. Their efficacy and safety have been tested in TS_COPD but not in BS-COPD. This trial will allow us to have a clinically and functionally characterization (using biological markers) of the BS-COPD phenotype and to compare those patients with those with the emphysema phenotype.

Hypothesis: Treatment with FF/V will be superior in preventing COPD exacerbations than the U/V combination in patients with COPD-asthma phenotype; while U/V will be superior than FF/V in patients with the emphysema phenotype.

General objective: To determine the exacerbations outcome (exacerbations free interval, exacerbations frequency, severe exacerbations that needed hospitalization frequency, exacerbations frequency according to absolute and percentage (>3%) blood eosinophils, exacerbations percentage for emphysema phenotype and COPD-asthma phenotype) in patients with COPD-asthma vs emphysema phenotype patients, treated with Fluticasone Furoate/Vilanterol 100/25 mcg/day vs Umeclidinium/Vilanterol 55/25 mcg/day, after 6 months of treatment.

Secondary objectives: To determine in both groups: (1) Pulmonary function change (FEV1, FVC and inspiratory capacity) (2) Impulse oscillometry resistance change (3) FeNO change (5) Quality of life change (CAT and Saint George) (6) Dyspnea change (mMRC, BDI y TDI) (7) Functional capacity change (6MWT distance). (8) To characterize and establish the frequency of the COPD-asthma phenotype in BS-COPD patients and emphysema-phenotype in TS-COPD patients.

Methods: Randomized double blind controlled clinical trial. Patients with at least one exacerbation in the last 12 months (confirmed by the prescription of antibiotic and/or oral steroid), and a smoking index > 10 packs/year or a biomass smoke exposition index > 100 hours/year. One hundred BS-COPD patients and one hundred TS-COPD patients will be included; both groups will be exposed to the two treatment options. Fifty patients from each group (BS-COPD and TS-COPD) will be assigned with FF/V and 50 from each group with U/V. Emphysema phenotype and air-trapping pattern will be determined with a CT image. All CTs will be assessed by a radiologist. Baseline DLco will also be correlated with the emphysema CT findings. Blood eosinophils, blood levels IgE, bronchodilator reversibility and baseline FeNO. Rate of exacerbations will be determined in both groups for a time period of 6 months. At the end of the study, the phenotype of each patient will be determined and treatment efficacy will be evaluated according to the phenotype. The sample size was chosen conventionally by considering that there are no other centers with a BS-COPD cohort. Treatment will be randomly assigned using a random numbers table. Safety evaluation includes severe adverse events (SAE) assessment (mainly pneumonia). During the informed consent signing visit (day -15), BS-COPD or TS-COPD diagnosis will be confirmed. There will be four in-clinic visits (baseline; +30 days; +90 days and +180 days) where the symptoms diary will be evaluated to determine the rate of exacerbations or other health resources use. Also, pulmonary function tests (spirometry pre and post-BD, IC) and functional capacity tests (6MWT) will be performed by each patient. Health related quality of life (SGRQ and CAT) and dyspnea (mMRC and BDI/TDI) questionnaires will also performed. There will be three telephonic visits (+60 days, +120 days, +210 days) where adverse events, concomitant medication, other health resources use and exacerbations since last visit will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 to 80 years
* Men and women (not fertile, not pregnant, or those with a effective birth control method)
* COPD diagnosis according to GOLD 2017 criteria with a FEV1 ≥ 30%
* Biomass smoke exposition index ≥ 100 hours/year or smoking index ≥ 10 packs/year,
* Patients with at least two exacerbations in the last 12 months (confirmed by the prescription of antibiotic and/or oral steroid)
* Patients with stable COPD (no exacerbations or respiratory infections in the 4 weeks prior inclusion).

Exclusion Criteria:

* Patients with allergies or intolerance to study medications
* Female patients on pregnancy, lactancy
* Patients with cancer diagnosis
* Patients with bronchiectasis, tuberculosis, recent COPD exacerbation, or any respiratory infection or cardiovascular anomaly that withholds the respiratory function test

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Exacerbations rate | baseline to 24 weeks
  moderate and severe exacerbations rate
Exacerbations free interval | Baseline to first exacerbation
  Exacerbations free interval

SECONDARY OUTCOMES:
Pulmonary function change | Change from Baseline at 4, 12 and 24 weeks
  Spirometry (FVC and FEV1) and inspiratory capacity
Impulse oscillometry resistance change | Change from baseline at 24 weeks
  R5, R20, DR5R20, Ax (percentage of expected in all values)
FeNO change | change from Baseline at 24 weeks
  ppb
Quality of life change | change from Baseline at 4, 12 and 24 weeks
  CAT
Dyspnea change | Change from Baseline at 4, 12 and 24 weeks
  mMRC
Functional capacity change | Change from Baseline at 4, 12 and 24 weeks
  6 minute walk test distance
SGRQ Quality of life change | Change from Baseline at 4, 12 and 24 weeks
  SGRQ

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Ramírez-Venegas, M.S., Principal Investigator — Instituto Nacional de Enfermedades Respiratorias
Locations (1):
- National Institute of Respiratory Diseases 'Ismael Cosío Villegas', Mexico City, Tlalpan, Mexico

REFERENCES:
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] Camp PG, Ramirez-Venegas A, Sansores RH, Alva LF, McDougall JE, Sin DD, Pare PD, Muller NL, Silva CI, Rojas CE, Coxson HO. COPD phenotypes in biomass smoke- versus tobacco smoke-exposed Mexican women. Eur Respir J. 2014 Mar;43(3):725-34. doi: 10.1183/09031936.00206112. Epub 2013 Oct 10. PMID 24114962
- [Background] Lopez Varela MV, Muino A, Perez Padilla R, Jardim JR, Talamo C, Montes de Oca M, Valdivia G, Pertuze J, Halbert R, Menezes AM; PLATINO Group. [Treatment of chronic obstructive pulmonary disease in 5 Latin American cities: the PLATINO study]. Arch Bronconeumol. 2008 Feb;44(2):58-64. doi: 10.1016/s1579-2129(08)60016-6. Spanish. PMID 18361870
- [Background] Caballero A, Torres-Duque CA, Jaramillo C, Bolivar F, Sanabria F, Osorio P, Orduz C, Guevara DP, Maldonado D. Prevalence of COPD in five Colombian cities situated at low, medium, and high altitude (PREPOCOL study). Chest. 2008 Feb;133(2):343-9. doi: 10.1378/chest.07-1361. Epub 2007 Oct 20. PMID 17951621
- [Background] Ramirez-Venegas A, Sansores RH, Quintana-Carrillo RH, Velazquez-Uncal M, Hernandez-Zenteno RJ, Sanchez-Romero C, Velazquez-Montero A, Flores-Trujillo F. FEV1 decline in patients with chronic obstructive pulmonary disease associated with biomass exposure. Am J Respir Crit Care Med. 2014 Nov 1;190(9):996-1002. doi: 10.1164/rccm.201404-0720OC. PMID 25172140
- [Background] Bruce N, Perez-Padilla R, Albalak R. Indoor air pollution in developing countries: a major environmental and public health challenge. Bull World Health Organ. 2000;78(9):1078-92. PMID 11019457
- [Background] Regalado J, Perez-Padilla R, Sansores R, Paramo Ramirez JI, Brauer M, Pare P, Vedal S. The effect of biomass burning on respiratory symptoms and lung function in rural Mexican women. Am J Respir Crit Care Med. 2006 Oct 15;174(8):901-5. doi: 10.1164/rccm.200503-479OC. Epub 2006 Jun 23. PMID 16799080
- [Background] Moran-Mendoza O, Perez-Padilla JR, Salazar-Flores M, Vazquez-Alfaro F. Wood smoke-associated lung disease: a clinical, functional, radiological and pathological description. Int J Tuberc Lung Dis. 2008 Sep;12(9):1092-8. PMID 18713510
- [Background] Rivera RM, Cosio MG, Ghezzo H, Salazar M, Perez-Padilla R. Comparison of lung morphology in COPD secondary to cigarette and biomass smoke. Int J Tuberc Lung Dis. 2008 Aug;12(8):972-7. PMID 18647460
- [Background] Usmani OS, Barnes PJ. Assessing and treating small airways disease in asthma and chronic obstructive pulmonary disease. Ann Med. 2012 Mar;44(2):146-56. doi: 10.3109/07853890.2011.585656. Epub 2011 Jun 17. PMID 21679101
- [Background] Vestbo J; TORCH Study Group. The TORCH (towards a revolution in COPD health) survival study protocol. Eur Respir J. 2004 Aug;24(2):206-10. doi: 10.1183/09031936.04.00120603. PMID 15332386
- [Background] Celli B, Decramer M, Kesten S, Liu D, Mehra S, Tashkin DP; UPLIFT Study Investigators. Mortality in the 4-year trial of tiotropium (UPLIFT) in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2009 Nov 15;180(10):948-55. doi: 10.1164/rccm.200906-0876OC. Epub 2009 Sep 3. PMID 19729663
- [Background] Bujarski S, Parulekar AD, Sharafkhaneh A, Hanania NA. The asthma COPD overlap syndrome (ACOS). Curr Allergy Asthma Rep. 2015 Mar;15(3):509. doi: 10.1007/s11882-014-0509-6. PMID 25712010
- [Background] Brzostek D, Kokot M. Asthma-chronic obstructive pulmonary disease overlap syndrome in Poland. Findings of an epidemiological study. Postepy Dermatol Alergol. 2014 Dec;31(6):372-9. doi: 10.5114/pdia.2014.47120. Epub 2014 Dec 3. PMID 25610352
- [Background] Al-Kassimi FA, Alhamad EH, Al-Hajjaj MS, Raddaoui E, Alzeer AH, Alboukai AA, Somily AM, Cal JG, Ibrahim AF, Shaik SA. Can computed tomography and carbon monoxide transfer coefficient diagnose an asthma-like phenotype in COPD? Respirology. 2017 Feb;22(2):322-328. doi: 10.1111/resp.12902. Epub 2016 Sep 13. PMID 27623733
- [Background] Golpe R, Sanjuan Lopez P, Cano Jimenez E, Castro Anon O, Perez de Llano LA. Distribution of clinical phenotypes in patients with chronic obstructive pulmonary disease caused by biomass and tobacco smoke. Arch Bronconeumol. 2014 Aug;50(8):318-24. doi: 10.1016/j.arbres.2013.12.013. Epub 2014 Feb 25. English, Spanish. PMID 24576449
- [Background] Wedzicha JA, Banerji D, Chapman KR, Vestbo J, Roche N, Ayers RT, Thach C, Fogel R, Patalano F, Vogelmeier CF; FLAME Investigators. Indacaterol-Glycopyrronium versus Salmeterol-Fluticasone for COPD. N Engl J Med. 2016 Jun 9;374(23):2222-34. doi: 10.1056/NEJMoa1516385. Epub 2016 May 15. PMID 27181606
- [Background] Zach JA, Newell JD Jr, Schroeder J, Murphy JR, Curran-Everett D, Hoffman EA, Westgate PM, Han MK, Silverman EK, Crapo JD, Lynch DA; COPDGene Investigators. Quantitative computed tomography of the lungs and airways in healthy nonsmoking adults. Invest Radiol. 2012 Oct;47(10):596-602. doi: 10.1097/RLI.0b013e318262292e. PMID 22836310
- [Background] Miravitlles M, Calle M, Soler-Cataluna JJ. Clinical phenotypes of COPD: identification, definition and implications for guidelines. Arch Bronconeumol. 2012 Mar;48(3):86-98. doi: 10.1016/j.arbres.2011.10.007. Epub 2011 Dec 22. English, Spanish. PMID 22196477
- [Background] Cosio BG, Soriano JB, Lopez-Campos JL, Calle-Rubio M, Soler-Cataluna JJ, de-Torres JP, Marin JM, Martinez-Gonzalez C, de Lucas P, Mir I, Peces-Barba G, Feu-Collado N, Solanes I, Alfageme I, Casanova C; CHAIN Study. Defining the Asthma-COPD Overlap Syndrome in a COPD Cohort. Chest. 2016 Jan;149(1):45-52. doi: 10.1378/chest.15-1055. Epub 2016 Jan 6. PMID 26291753